CLINICAL TRIAL: NCT04436146
Title: The Effect of Laryngeal Manual Therapy as a Management of Globus(Sensation of a Lump in the Throat )- COMPARATIVE PROSPECTIVE STUDY
Brief Title: The Effect of Laryngeal Manual Therapy as a Management of Globus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Paker Miki, MD, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMC-20-0014
Record Dates: First submitted 2020-06-16; First posted 2020-06-17 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Globus
MeSH Terms: conditions — Globus Sensation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laryngeal manual therapies (Other): The laryngeal manual therapy incorporates massaging the laryngeal muscles thus reducing excessive tension in the laryngeal and perilaryngeal musculature in patients with globus .
  Interventions: Other: laryngeal manual therapies

INTERVENTIONS:
Other: laryngeal manual therapies — The laryngeal manual therapy incorporates massaging the laryngeal muscles thus reducing excessive tension in the laryngeal and perilaryngeal musculature in patients with globus .

SUMMARY:
The purpose of this study is to assess the effect of laryngeal manual therapies in the treatment of globus (sensation of a lump in the throat).

DETAILED DESCRIPTION:
This is a prospective study that include patients who met the inclusion criteria.

Data collection includes patients age,gender,clinical manifistations,laboratory parameters and treatment.

An endoscopic examination will be done by an expert Otolaryngologist. for each patients we will perform one session of laryngeal manual massage therapy by an expert in the field .

ELIGIBILITY:
Inclusion Criteria:

* patients more than 18 years old
* male and females
* patients complaning from Globus without an organic cause
* patients who underwent throat endoscopy and was normal.
* Patients who received conventional drug therapy without benefit.
* Globus complaints more than two months .

Exclusion Criteria:

* below 18
* Patients diagnosed with reflux(as a cause to globus)
* Patients who considered at high risk of reflux according to REFLUX SYMPTOM INDEX (RSI) more than 13
* patients who diagnosed with reflux and improved after anti-reflux manegment .
* patients with laryngeal disease/finding that can explain the globus.
* patients with organic cause that can explain the globus .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Change From symptomatic to asymptomatic patient | baseline and week 1
  after one therapy session we will evaluate the effect of the therapy on the patients .

CONTACTS AND LOCATIONS:
Overall Officials: Miki Paker, MD, Principal Investigator — HaEmek Medical Center, Israel
Locations (1):
- Haemek Medical Center, Afula, Israel